CLINICAL TRIAL: NCT05575401
Title: Post-operative Outcomes of Tonsillectomy With Lateral Pharyngoplasty Versus Tonsillectomy Alone in Children: a Randomized Controlled Trial
Brief Title: Lateral Pharyngoplasty Outcomes in Children Undergoing Tonsillectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5210282
Record Dates: First submitted 2022-10-07; First posted 2022-10-12 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Sleep-Disordered Breathing; Sleep Apnea Syndromes in Children; Sleep Apnea, Obstructive; Tonsillitis; Tonsillar Hypertrophy; Tonsil Stone; Tonsil Disease
Keywords: Tonsillectomy; Post-tonsillectomy hemorrhage; Post-tonsillectomy complication; Lateral pharyngoplasty
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Tonsillitis; tonsillolith | interventions — Tonsillectomy

STUDY DESIGN:
Intervention Model Description: Participants ages 3-17 years undergoing tonsillectomy for any reason will be randomized to either undergo tonsillectomy +/- adenoidectomy (standard of care practice) or tonsillectomy +/- adenoidectomy with lateral pharyngoplasty (research intervention). Parents of participants in both arms will be given post-operative worksheets to document pain scores, pain medication administration, estimates of daily per os intake, and any complications.
Who Masked: Participant
Masking Description: At the beginning of the study, each surgeon will receive an 80-item numbered list for which a random generator has been used to assign lateral pharyngoplasty or no lateral pharyngoplasty to each study participant. Each participant recruited for the study will undergo the correlating procedure at the time of surgery. Thus, the surgeon is necessarily not blinded, but the participant and parents would be blinded, and informed consent for the procedure would be for tonsillectomy +/- adenoidectomy, possible lateral pharyngoplasty.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tonsillectomy +/- adenoidectomy (Active Comparator): Participants will undergo extracapsular tonsillectomy +/- adenoidectomy.
  Interventions: Procedure: Tonsillectomy
- Tonsillectomy +/- adenoidectomy with lateral pharyngoplasty (Experimental): Participants will undergo extracapsular tonsillectomy +/- adenoidectomy and lateral pharyngoplasty.
  Interventions: Procedure: Lateral pharyngoplasty; Procedure: Tonsillectomy

INTERVENTIONS:
Procedure: Lateral pharyngoplasty — Two figure-of-8 sutures using 3-0 vicryl are used to approximate the anterior and posterior tonsillar pillars and reconstruct the continuous mucosal covering of the lateral pharyngeal walls.
  Arms: Tonsillectomy +/- adenoidectomy with lateral pharyngoplasty
Procedure: Tonsillectomy — Extracapsular tonsillectomy

SUMMARY:
The goal of this treatment study is to determine if doing lateral pharyngoplasty with tonsillectomy is better for children than doing tonsillectomy alone. The main questions it aims to answer are:

* Do children experience less pain after surgery when lateral pharyngoplasty is performed with tonsillectomy compared to tonsillectomy alone?
* Do children eat/drink better when lateral pharyngoplasty is performed with tonsillectomy compared to tonsillectomy alone?
* Is there a lower risk of bleeding after tonsillectomy when lateral pharyngoplasty is performed? Researchers will compare children undergoing tonsillectomy and lateral pharyngoplasty with children undergoing tonsillectomy alone to see if the participants experience less pain, better oral intake, and less bleeding complications after surgery. Parents of participants will be asked to record pain scores and pain medications given, approximate amounts of daily oral intake, and any complications after surgery.

DETAILED DESCRIPTION:
This is a randomized controlled trial to elucidate the benefits of performing lateral pharyngoplasty with tonsillectomy and encourage its use as a standard of care procedure. Participants will be randomized to receive either tonsillectomy +/- adenoidectomy or tonsillectomy +/- adenoidectomy with lateral pharyngoplasty (research intervention), with lateral pharyngoplasty referring to the placement two figure-of-8 sutures with 3-0 vicryl to reapproximate the anterior and posterior tonsillar pillars on each side. The investigators' hypothesis is that participants undergoing lateral pharyngoplasty will experience less pain, lower post-tonsillectomy hemorrhage rate, and a faster return to normal oral intake than participants undergoing tonsillectomy alone.

ELIGIBILITY:
Inclusion Criteria:

* Participants ages 3-17 years of age undergoing tonsillectomy +/- adenoidectomy at Loma Linda University Health

Exclusion Criteria:

* Subjects with congenital syndromes and/or developmental delay
* Subjects with cancer
* Subjects with gastrostomy tube use or dependence
* Subjects undergoing intracapsular tonsillectomy

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2023-05-17 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Level of post-operative pain | Change between baseline (immediately post-op) through 6 weeks after surgery
  Will use the Wong-Baker FACES pain scale, which shows a series of faces ranging from a happy face at 0 (representing no pain) to a crying face at 10 (representing the worst pain imaginable). Parent/caregiver will document the pain score and pain medication administrations/duration of use.
Number of participants with post-tonsillectomy hemorrhage requiring surgical intervention | Change between baseline (immediately post-op) through 6 weeks after surgery
  Count of subjects who undergo control of post-tonsillectomy hemorrhage in the operating room
Number of participants with post-tonsillectomy hemorrhage not requiring surgical intervention | Change between baseline (immediately post-op) through 6 weeks after surgery
  Count of subject/caregiver reports or presentations to a healthcare facility due to a post-tonsillectomy hemorrhage event that does not require control of hemorrhage in the operating room

SECONDARY OUTCOMES:
Post-operative duration (in days) to normal oral intake | Change between baseline (immediately post-op) through 6 weeks after surgery
  Parent/caregiver's will estimate the participant's daily soft diet oral intake as a percentage of perceived baseline/normal

OTHER OUTCOMES:
Number of participants requiring intravenous fluid administration for dehydration | Change between baseline (immediately post-op) through 6 weeks after surgery
  Presentation to healthcare facility due to lack of/perceived inadequate oral intake or decreased urination requiring intravenous fluid administration

CONTACTS AND LOCATIONS:
Overall Officials: Tsungju O-Lee, MD, Principal Investigator — Loma Linda University Health
Locations (4):
- United States (4):
  - Loma Linda University Professional Building - Murrieta, Murrieta, California
  - Loma Linda University ENT/Head & Neck Surgery, Riverside, California
  - Pediatric Ear, Nose, and Throat Surgery and Audiology, San Bernardino, California
  - SAC Health - ENT Clinic, San Bernardino, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Genc E, Hanci D, Ergin NT, Dal T. Can mucosal sealing reduce tonsillectomy pain? Int J Pediatr Otorhinolaryngol. 2006 Apr;70(4):725-30. doi: 10.1016/j.ijporl.2005.12.005. Epub 2006 Jan 18. PMID 16414127
- [Background] Kim JS, Kim BG, Kim DH, Hwang SH. Efficacy of pillar suture for post-tonsillectomy morbidity in children: a meta-analysis. Braz J Otorhinolaryngol. 2021 Sep-Oct;87(5):583-590. doi: 10.1016/j.bjorl.2019.12.007. Epub 2020 Jan 25. PMID 32057680
- [Background] Ramjettan S, Singh B. Are sutured faucial pillars really an advantage in tonsillectomy? S Afr J Surg. 1996 Nov;34(4):189-91. PMID 9015944
- [Background] Shu Y, Yao HB, Yang DZ, Wang B. Postoperative characteristics of combined pharyngoplasty and tonsillectomy versus tonsillectomy in children with obstructive sleep apnea syndrome. Arch Argent Pediatr. 2018 Oct 1;116(5):316-321. doi: 10.5546/aap.2018.eng.316. English, Spanish. PMID 30204981
- [Background] Wulu JA, Chua M, Levi JR. Does suturing tonsil pillars post-tonsillectomy reduce postoperative hemorrhage?: A literature review. Int J Pediatr Otorhinolaryngol. 2019 Feb;117:204-209. doi: 10.1016/j.ijporl.2018.12.003. Epub 2018 Dec 4. PMID 30611028